CLINICAL TRIAL: NCT07170475
Title: A Phase Ib Trial of Combined Febuxostat and Inosine Therapy in Patients With Parkinson's Disease
Acronym: iFRESH-PD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujita Health University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FU-PD-i01
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson Disease; Febuxostat; Inosine; Hypoxanthine; Combination Therapy; Safety Study
MeSH Terms: conditions — Parkinson Disease | interventions — Febuxostat; Inosine

STUDY DESIGN:
Intervention Model Description: Participants are randomized in parallel to one of four dose-combination groups and receive their assigned regimen twice daily for 12 weeks. Dosing is open-label, with febuxostat co-administered with inosine each morning and evening. Safety and pharmacodynamic blood measures are collected at baseline and at weeks 4, 8, and 12.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - Febuxostat + Inosine （Dose Level 1) (Experimental): Participants receive febuxostat and inosine (Dose Level 1) orally, twice daily (once in the morning and once in the evening) for 12 weeks.
  Interventions: Drug: Febuxostat; Drug: Inosine
- Group 2 - Febuxostat + Inosine (Dose Level 2) (Experimental): Participants receive febuxostat and inosine (Dose Level 2) orally, twice daily (once in the morning and once in the evening) for 12 weeks.
  Interventions: Drug: Febuxostat; Drug: Inosine
- Group 3 - Febuxostat + Inosine (Dose Level 3) (Experimental): Participants receive febuxostat and inosine (Dose Level 3) orally, twice daily (once in the morning and once in the evening) for 12 weeks.
  Interventions: Drug: Febuxostat; Drug: Inosine
- Group 4 - Febuxostat + Inosine (Dose Level 4) (Experimental): Participants receive febuxostat and inosine (Dose level 4) orally, twice daily (once in the morning and once in the evening) for 12 weeks.
  Interventions: Drug: Febuxostat; Drug: Inosine

INTERVENTIONS:
Drug: Febuxostat — Febuxostat tablets (per randomized assignment), administered orally twice daily (once in the morning and once in the evening) for 12 weeks.
Drug: Inosine — Inosine tablets (per randomized assignment), administered orally twice daily (once in the morning and once in the evening) for 12 weeks.

SUMMARY:
This study will test the safety of twice-daily oral dosing of combined febuxostat and inosine in 24 patients with Parkinson's disease. Participants will receive one of the four regimens, taken twice daily for 12 weeks:

Who can join: Adults with early-stage Parkinson's disease on stable medication regimens.

What participants do:

* Take their assigned dose twice daily (morning and evening) for 12 weeks.
* Visit the clinic at baseline and weeks 4, 8, and 12 for blood tests (including hypoxanthine), exams, and questionnaires.
* Keep a simple diary of any side effects or changes in daily activities.

Risks and benefits: Possible side effects include mild gastrointestinal upset, headache, or elevated uric acid levels. While direct benefit is not guaranteed, this safety data will inform future Parkinson's disease treatments.

Learn more: Contact [site-specific contact info] for details on eligibility and enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide voluntary written informed consent.
2. Receiving stable Parkinson's disease medication (no changes in type or dose) for at least 3 months before enrollment.
3. Age 18 to 80 years at the time of consent.
4. Diagnosed with Parkinson's disease by a specialist according to MDS-PD diagnostic criteria, and at pre-enrollment screening, all of the following are met:

   1. Hoehn-Yahr stage (ON state) 1 to 3
   2. MDS-UPDRS Part III (ON state) score 10 to 35
   3. Mini-Mental State Examination (MMSE) score ≥ 24

Exclusion Criteria:

1. Requires almost total assistance in daily life and is unable to walk or stand unaided.
2. Currently taking azathioprine, mercaptopurine hydrate, vidarabine, didanosine, or rosuvastatin.
3. Used febuxostat, allopurinol, or topiroxostat within 3 months before study start.
4. Taking any supplement containing inosine.
5. Started any new Parkinson's disease medication or therapy within 3 months before enrollment.
6. Serum creatinine >1.5× upper limit of normal (ULN), or AST (GOT) or ALT (GPT) >2× ULN at screening.
7. History of surgical treatment for Parkinson's disease.
8. History of or comorbid hypersensitivity/allergy to any ingredient of the investigational drugs.
9. Participation in another clinical trial involving an unapproved drug within 30 days before consent, or currently enrolled in another interventional study.
10. Pregnant or breastfeeding, or unwilling/unable to use reliable contraception during the study period.
11. Positive test at screening for HIV, HBV, HTLV-1, or syphilis; **HCV antibody-positive with undetectable HCV RNA** is allowed.
12. Unable to take the investigational drugs orally without changing the dosage form.
13. Gastrointestinal disease or prior GI surgery that may affect drug absorption, as judged by the investigator.
14. Psychiatric disorder or symptoms that interfere with daily life and make study participation difficult.
15. Unable to complete assessments or questionnaires independently.
16. Any other condition that, in the investigator's judgment, would make participation unsafe or inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma hypoxanthine concentration from baseline to Week 12 | 12 weeks
  The difference in plasma hypoxanthine level (µmol/L) between pre-dose at Day 0 and Week 12 visit.

SECONDARY OUTCOMES:
Change in plasma hypoxanthine concentration from baseline to Week 4 | 4 weeks
  The difference in plasma hypoxanthine level between pre-dose at Day 0 and Week 4 visit.
Change in cerebrospinal fluid (CSF) hypoxanthine concentration from baseline to Week 12 | 12 weeks
  The difference in CSF hypoxanthine level between the pre-dose at Day 0 and the Week 12 visit.
Change in MDS-UPDRS Part III score from baseline to Week 12 | 12 weeks
  The difference in Movement Disorder Society-Unified Parkinson's Disease Rating Scale motor examination (ON state) score between Day 0 and Week 12.
Change in Mini-Mental State Examination (MMSE) score from baseline to Week 12 | 12 weeks
  The difference in MMSE score between Day 0 and Week 12.
Change in Geriatric Depression Scale-15 (GDS-15) score from baseline to Week 12 | 12 weeks
  The difference in GDS-15 score between Day 0 and Week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujita Health University, Toyoake, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including the dataset and data dictionary) and the whole study protocol will be made available to qualified researchers beginning 6 months after publication and ending 3 years after publication. Requests should be directed to the corresponding author, Dr. Hirohisa Watanabe (email: hirohisa.watanabe@fujita-hu.ac.jp), with a research proposal and data use agreement.
  IPD Sharing Time Frame: Available 6 months to 3 years after publication. IPD Sharing Access Criteria: Qualified researchers with IRB/ethics approval and a signed data use agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available 6 months to 3 years after publication of the primary results.
Access Criteria: Qualified researchers who have obtained approval from their institutional review board or ethics committee and who sign a data use agreement with the study sponsor may request access to de-identified individual participant data, the full study protocol, statistical analysis plan, informed consent form, and analytic code. Requests should be submitted via email to the corresponding author, Dr. Hirohisa Watanabe (hirohisa.watanabe@fujita-hu.ac.jp), and include a brief research proposal and evidence of IRB/ethics approval.
URL: https://jrct.mhlw.go.jp/en-latest-detail/jRCT2041250029

REFERENCES:
- [Background] Kamatani N, Hashimoto M, Sakurai K, Gokita K, Yoshihara J, Sekine M, Mochii M, Fukuuchi T, Yamaoka N, Kaneko K. Clinical studies on changes in purine compounds in blood and urine by the simultaneous administration of febuxostat and inosine, or by single administration of each. Gout and Nucleic Acid Metabolism. 2017;41 (2): 171-181.
- [Background] Kamatani N, Kushiyama A, Toyo-Oka L, Toyo-Oka T. Treatment of two mitochondrial disease patients with a combination of febuxostat and inosine that enhances cellular ATP. J Hum Genet. 2019 Apr;64(4):351-353. doi: 10.1038/s10038-018-0558-0. Epub 2019 Jan 10. PMID 30631120
- [Background] Johnson TA, Jinnah HA, Kamatani N. Shortage of Cellular ATP as a Cause of Diseases and Strategies to Enhance ATP. Front Pharmacol. 2019 Feb 19;10:98. doi: 10.3389/fphar.2019.00098. eCollection 2019. PMID 30837873
- [Background] Shima S, Mizutani Y, Yoshimoto J, Maeda Y, Ohdake R, Nagao R, Maeda T, Higashi A, Ueda A, Ito M, Mutoh T, Watanabe H. Uric acid and alterations of purine recycling disorders in Parkinson's disease: a cross-sectional study. NPJ Parkinsons Dis. 2024 Sep 9;10(1):170. doi: 10.1038/s41531-024-00785-0. PMID 39251680
- [Background] Watanabe H, Hattori T, Kume A, Misu K, Ito T, Koike Y, Johnson TA, Kamitsuji S, Kamatani N, Sobue G. Improved Parkinsons disease motor score in a single-arm open-label trial of febuxostat and inosine. Medicine (Baltimore). 2020 Aug 28;99(35):e21576. doi: 10.1097/MD.0000000000021576. PMID 32871874